CLINICAL TRIAL: NCT00531141
Title: Reproducibility of Retinal Thickness Measurements by Optical Coherence Tomography in Age-Related Macular Degeneration The OCT in AMD Study
Brief Title: The Optical Coherence Tomography in Age-Related Macular Degeneration Study: The OCT in AMD Study
Status: Completed | Type: Observational
Sponsor: The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery (Other)
Responsible Party: Susanne Binder Prof, The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery
Other Study IDs: EK 07-078-VK
Record Dates: First submitted 2007-09-15; First posted 2007-09-18 (Estimated); Last update posted 2009-06-24 (Estimated); Status verified 2009-06

CONDITIONS: Macular Degeneration
Keywords: age-related macular degeneration; optical coherence tomography; retinal thickness; exudative age-related macular degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- A: examination twice by examiner 1
  Interventions: Other: examination only
- B: examination first by examiner 1 thereafter by examiner 2
  Interventions: Other: examination only
- C: examination first by examiner 2 thereafter by examiner 1
  Interventions: Other: examination only
- D: examination performed twice by examiner 2
  Interventions: Other: examination only

INTERVENTIONS:
Other: examination only — OCT performed twice

SUMMARY:
The Optical Coherence Tomography (OCT) is a non-contact, non invasive method to examine the retina by providing cross-sectional scans through the retina. Measurements of the retinal thickness based on automatically set border lines created by threshold algorithm provide information concerning the amount of intraretinal fluid and activity of the lesion. In this study the reproducibility of retinal thickness measurements in patients suffering from age-related macular degeneration performed by two independent examiners of two examinations of the same day but performed in a time interval of at least two hours should be evaluated. Using the macular thickness program of stratus OCT, 6 radial lines through the center of the foveal avascular zone are performed, Differences between the first and second measurement will be investigated by a 95% confidence interval, a Bland-Altman plot (with corresponding regression analysis) and a random effect model with time, examiner and diagnosis as fixed factors. Although threshold algorithm failures and fixation problems are common in age-related macular degeneration evidence of reproducibility and repeatability of maximum retinal thickness is expected.

ELIGIBILITY:
Inclusion Criteria:

* Age over 50 years
* Age related macular degeneration

Exclusion Criteria:

* Macular pathologies other than age related macular degeneration (diabetic maculopathy, macular pucker, macular hole,
* Visualization of the macula not possible (dens cataract, vitreous haemorrhage)
* Not consented patients

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2007-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ilse Krebs, MD, Principal Investigator — Rudolf Foundation Clinic
Locations (1):
- Ludwig Boltzmann Institute for Retinology and Biomicroscopic Lasersurgery, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Krebs I, Hagen S, Brannath W, Haas P, Womastek I, de Salvo G, Ansari-Shahrezaei S, Binder S. Repeatability and reproducibility of retinal thickness measurements by optical coherence tomography in age-related macular degeneration. Ophthalmology. 2010 Aug;117(8):1577-84. doi: 10.1016/j.ophtha.2010.04.032. Epub 2010 Jun 16. PMID 20557937